CLINICAL TRIAL: NCT04162860
Title: Preemptive Endoluminal Negative Pressure Therapy at the Anastomotic Site in Minimally Invasive Transthoracic Esophagectomy - An International Multicenter Randomized Controlled Trial
Brief Title: Preemptive Endoluminal Negative Pressure in Minimally Invasive Transthoracic Esophagectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Christian Gutschow, Professor, Head of upper gastrointestinal unit, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-00562
Record Dates: First submitted 2019-07-11; First posted 2019-11-14 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Esophageal Cancer; Surgery--Complications; Leak, Anastomotic
MeSH Terms: conditions — Esophageal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimally invasive esophagectomy with preemptive ENP (Experimental): Patients will undergo a standard total minimally invasive transthoracic Ivor Lewis esophagectomy with preemptive ENP. After completion of the esophago-gastric anastomosis, an Eso-SPONGE® system will be inserted via an intraoperative gastroscopy. ENP will be carried out upon completion of the esophago-gastrostomy, but no later than 12 hours after the surgical intervention. Postoperatively, secretions are then continuously evacuated using a suction pump generating a negative pressure between 75 and 100 mmHg. ENP will remain for 4 days and will be monitored with clinical parameters.
  Interventions: Device: Eso-SPONGE® device
- Standard minimally invasive esophagectomy (No Intervention): Patients in the control group will undergo a standard minimally invasive transthoracic Ivor Lewis esophagectomy without preemptive ENP.

INTERVENTIONS:
Device: Eso-SPONGE® device — Preemptive ENP therapy will be carried out with either an Eso-SPONGE® device system (Eso-SPONGE®, B. Braun Melsungen AG, Melsungen, Germany). Eso-SPONGE® consists of an open-pored polyurethane foam fitted to a gastric tube. Secretions are then continuously evacuated using a suction pump generating a negative pressure between 75 and 100 mmHg.
  Arms: minimally invasive esophagectomy with preemptive ENP

SUMMARY:
The primary objective of the preSponge randomized controlled trial (RCT) will be to assess the potential protective effects of preemptive endoscopic negative pressure therapy (ENP) on postoperative morbidity in high-risk patients undergoing total minimally invasive transthoracic esophagectomy with gastric pull-up reconstruction and high intrathoracic anastomosis (thoracoscopic and laparoscopic Ivor Lewis esophagectomy).

ELIGIBILITY:
Inclusion Criteria:

We will include adult patients (≥18 years of age) with resectable esophageal cancer (adenocarcinoma or squamous cell carcinoma) with high risk for anastomotic leakage (AL) who provided informed consent and are scheduled for minimally invasive transthoracic Ivor Lewis esophagectomy. Robotic-assisted procedures will also be included.

Patients considered at high risk for AL must have at least one of the following risk factors:

* American Society of Anesthesiologists Classification (ASA) score >2
* Diabetes (insulin dependent or HbA1c ≥ 6.5%)
* Chronic pulmonary disease (first second of forced expiration (FEV1)/Forced volume vital capacity (FVC) ratio ≤ 70%)
* Heart failure (left ventricular ejection fraction (LVEF) <55%)
* Preexisting cardiac arrhythmia (pacemaker or paroxysmal supraventricular tachyarrhythmia)
* Chronic kidney disease stage 4-5 (glomerular filtration rate (GFR) < 30ml/min/1.73 m2)
* Chronic liver disease with treated portal hypertension (porto-caval pressure gradient ≥5-≤10mmHg, including patients with transjugular intrahepatic portosystemic shunt (TIPS))
* Previous radiotherapy or chemo-radiation ≥50Gray (Gy) (salvage esophagectomy)

Alternatively, patients must have at least two of the following risk factors:

* Arteriosclerosis score 2 according to van Rossum et al.13 (aorta and coeliac axis)
* Malnutrition (Body mass index (BMI) ≤ 18.5kg/m2)
* Obesity (BMI ≥ 35kg/m2)
* Heart failure with preserved ejection fraction (LVEF >55%)
* Active or former smoking
* Age > 65 years
* World health Organisation (WHO)/Zubrodt score > 1
* chronic kidney disease stage 2-3 (GFR 30-89 ml/min/1.73 m2)
* chronic liver disease without portal hypertension (porto-caval pressure gradient ≤5mmHg)

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, or dementia.
* Patients younger than 18 years
* Patients undergoing esophagectomy for benign disease or for malignancy other than adenocarcinoma or squamous cell carcinoma
* Patients scheduled for other technical variants of esophagectomy, such as open, hybrid, or transhiatal procedures (intraoperative conversions to open access surgery will not be excluded)
* Chronic liver disease with portal hypertension (porto-caval pressure gradient >10mmHg)
* Distant organ metastasis (cM+)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay until "fit-for-discharge" criteria are reached | 90-days postoperatively
  * The patients' oral/enteral nutritional requirements are met by oral intake of at least liquids with optional supplementary nutrition via jejunal feeding tube.
  * The patient should have passed flatus.
  * The patient does not require oxygen during mobilisation (short walk or climbing stairs) or at rest.
  * Central venous catheters should be removed before discharge (unless present preoperatively).
  * Adequate analgesia at rest and during mobilisation (pain score <4 on a scale from 0 to 10) is achieved using both oral opioid and non-opioid analgesics.
  * All vital signs should be normal unless abnormal preoperatively.
  * Inflammatory parameters (white cell count, C-reactive protein) should be trending down and close to normal.
  * There should be adequate support after discharge (assistance by family, ambulatory nursing, or rehabilitation facility).

SECONDARY OUTCOMES:
Postoperative Complications | 90-days postoperatively
  Assessment of postoperative complications according to Clavien-Dindo
Postoperative Complications | 90-days postoperatively
  Hospital readmissions
Postoperative Complications | 90-days postoperatively
  Anastomotic stricture

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gutschow, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Muller PC, Vetter D, Kapp JR, Gubler C, Morell B, Raptis DA, Gutschow CA. Pre-Emptive Endoluminal Negative Pressure Therapy at the Anastomotic Site in Minimally Invasive Transthoracic Esophagectomy (the preSPONGE Trial): Study Protocol for a Multicenter Randomized Controlled Trial. Int J Surg Protoc. 2021 Mar 18;25(1):7-15. doi: 10.29337/ijsp.24. PMID 34013139